CLINICAL TRIAL: NCT04556240
Title: RECORD-VP: Real-time Evaluation of Cardiac Outpatient Recording Device With VitalPatch RTM
Status: Withdrawn | Type: Observational
Why Stopped: Study withdrawn due to COVID endemic
Sponsor: VitalConnect Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-323
Record Dates: First submitted 2020-09-02; First posted 2020-09-21 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Arrhythmias, Cardiac
Keywords: Arrhythmias; Real-time Monitoring; Mobile Cardiac Telemetry; VitalPatch; Independent Diagnostic Testing Facility
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: VitalConnect Platform — The VitalConnect Platform is a wireless remote monitoring system intended for use by healthcare professionals for continuous collection of physiological and irregular heart rhythm data in home and healthcare settings. This includes heart rate, electrocardiogram (ECG), heart rate variability (R-R interval), breathing rate, arrhythmia detection, body temperature, skin temperature, activity (including step count), and posture (body position relative to gravity including fall). Data is transmitted wirelessly to a central location where it is stored for analysis. The VitalConnect Platform can be configured by authorized persons to notify healthcare professionals when physiological data falls outside selected parameters

SUMMARY:
The primary purpose of this study is to evaluate performance and safety of the VitalConnect Platform when used for mobile cardiac telemetry (MCT) or as an independent diagnostic testing facility (IDTF) system during activities of daily living by subjects 18 years or older who have been recommended MCT by their care provider.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. If recommended mobile cardiac telemetry (MCT) by the care provider
3. If instructed, be willing to record information such as daily activities and symptoms
4. Able to speak, read, and write English.

Exclusion Criteria:

1. Have extensive skin changes/diseases that preclude wearing the required number of devices on normal skin at the proposed wear sites;
2. Have a known allergy to medical adhesives;
3. Have any potentially life-threatening condition that (for example ventricular tachycardia or ventricular fibrillation), in the opinion of the Investigator, would interfere with their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of up to five-hundred (500) non-randomized subjects who have been recommended mobile cardiac telemetry by their care provider.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Successfully detect heart rhythm of the study subjects using VitalConnect platform as a mobile cardiac telemetry unit | Each patient will be monitored for up-to 30 days
  Monitor the heart rhythm of the study subjects initially for up to 24 hours and if the monitoring finds the issue that the doctor is looking for, the monitoring will be stopped. In most of the cases, the monitoring can continue for up to 30 days for each study subject

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Sheehan, MD, Principal Investigator — VitalConnect Inc.
Locations (1):
- Site 1, Chevy Chase, Maryland, United States

IPD SHARING:
Plan to Share IPD: No